CLINICAL TRIAL: NCT02761135
Title: Does End-fire Technique Increase Detection Rate of Prostate Cancer at First Re-biopsy Compared to Side-fire Technique, in Investigating a Raised Prostatic Specific Antigen (PSA)?
Brief Title: Does End-fire Technique Increase Detection Rate of Prostate Cancer at First Re-biopsy Compared to Side-fire Technique?
Status: Completed | Type: Observational
Sponsor: Kronoberg County Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: Endfirestudie
Record Dates: First submitted 2015-05-21; First posted 2016-05-04 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Biopsy technique; Transrectal ultrasonography probe; Side-fire; Prostate cancer; End-fire
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy cores from prostate.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Side-fire: Using side-fire technique during transrectal ultrasound.
- End-fire: Using end-fire technique during transrectal ultrasound.

SUMMARY:
Prostate cancer is the most common cancer among men in Sweden. During investigation of suspected cancer transrectal ultrasound with needle biopsies from prostate leeds to diagnosis.

The most common technique today is side-fire where the needle enter the prostate in angle from the probe. In end-fire technique the needle enters the prostate at tip of probe without angle. The difference in techniques side-fire vs. end-fire affects the possibility to reach the ventral and apical aspects of prostate.

Today´s standard is at least five cores from each side of the prostate at first biopsy. If first sample is negative there will usually be another urological exam and a first re-biopsy.

The study aim to compare these two methods in cancer detection. The investigators' hypothesis is that when using end-fire technique at first re-biopsy, investigators find more cancers compared to side-fire.

Patients are prospectively randomized into two groups, both assessing 12 core biopsies according to study protocol.

Primary endpoint is cancer detection. Data will be collected about patient age, PSA-level, prostate size, digital rectal exam, hypoechogenic zones and length of cancers.

ELIGIBILITY:
Inclusion Criteria:

* first re-biopsy
* PSA over 3ng/ml
* T1c to T2a palpatory finding

Exclusion Criteria:

* prostate cancer
* T2b or more advanced cancer
* more than one previous biopsy done

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men admitted to Urological reception in Vaxjo and Ljungby for a first-time re-biopsy for investigating prostate cancer.
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2011-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cancer detection | Study inclusion continues until 400 patients is included. Estimated time frame from study start 5 years.
  After finished study inclusion, data will be analyzed and presented within 12-18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Ortegren, Principal Investigator — Section of Urology, Department of Surgery, Växjö County Hospital, Växjö, Sweden
Locations (1):
- Section of Urology, Department of surgery, Regional Hospital Växjö, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ortegren J, Holmberg JT, Lekas E, Mana S, Martensson S, Richthoff J, Sundqvist P, Kjolhede H, Bratt O, Liedberg F. A randomised trial comparing two protocols for transrectal prostate repeat biopsy: six lateral posterior plus six anterior cores versus a standard posterior 12-core biopsy. Scand J Urol. 2019 Aug;53(4):217-221. doi: 10.1080/21681805.2019.1628102. Epub 2019 Jun 17. PMID 31204873